CLINICAL TRIAL: NCT01002105
Title: Baclofen as Add-On to Standard Treatment of Alcohol- Dependent Patients and Its Effect on Quality of Life, Clinical and Psychosocial Features: A 12-Week Double-Blind Randomized Controlled Trial
Brief Title: Baclofen as Add-On to Standard Treatment of Alcohol- Dependent Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sha'ar Menashe Mental Health Center (Other)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Principal Investigator, Alexander Grinshpoon, Dr. Alexander Grinshpoon, Sha'ar Menashe Mental Health Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AGRIN4CTIL
Record Dates: First submitted 2009-10-19; First posted 2009-10-27 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-11

CONDITIONS: Alcohol Dependence
Keywords: Baclofen; Alcohol; Baclofen as add-on to standard treatment of alcohol
MeSH Terms: conditions — Alcoholism | interventions — Baclofen; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baclofen (Experimental): The study was a double-blind, placebo-controlled, randomized trial comparing 50 mg/day of baclofen to placebo over 12 weeks, in addition to a low-intensity psychosocial intervention program, with 26-week and 52-week follow-up observations.
  Interventions: Drug: Baclofen
- Psychosocial intervention (Other): Intervention of the addition of placebo to low-intensity psychosocial intervention program. This was the control group
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Baclofen — Baclofen 50mg per day for 12 weeks and psychosocial intervention
  Arms: Baclofen
Other: Control group — psychosocial intervention and placebo for 12 weeks
  Other Names: Placebo group
  Arms: Psychosocial intervention

SUMMARY:
This is a study of Baclofen as an add-on to standard treatment for alcohol-dependent patients.

DETAILED DESCRIPTION:
Double-blind, placebo-controlled, randomized trial comparing 50 mg/day of baclofen to placebo over 12 weeks, in addition to a low-intensity psychosocial intervention program, with 26-week and 52-week follow-up observations. The percentages of heavy drinking days and abstinent days were the primary outcome measures, and craving; distress and depression levels; self-efficacy; social support from family, friends and significant others; and health-related quality of life (HRQL) were secondary outcomes. Tolerability was also examined.

ELIGIBILITY:
Inclusion Criteria:

1. ICD-10 diagnosis of alcohol dependence (World Health Organization, 1993);
2. Seeking treatment with the aim to stop alcohol consumption;
3. Age ranging from 18 to 60 years;
4. Last alcohol intake reported in the 24 h preceding observation;
5. Presence of a referred family member;
6. Written informed consent provision.

Exclusion Criteria:.

1. Serious hepatic, kidney, lung, neurological and cardiovascular, diseases);
2. Suicide risk, acute psychosis, severe depression, organic brain syndromes;
3. Dependence on psychoactive substances other than nicotine.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M Ponizovsky, MD, PhD, Study Director — Ministry of health, State of Israel
Locations (1):
- Alexander Grinshpoon, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1/1/2009 - 31 /12/2010, 75 patients recruited from 15 outpatient centers. Of 75, 4 refused and 7 did not meet the inclusion criteria and 64 patients (48 male and 16 female) were randomly assigned either to baclofen (N=32) or placebo (N=32) in a double-bli
Groups:
- Baclofen: The study was a double-blind, placebo-controlled, randomized trial comparing 50 mg/day of baclofen to placebo over 12 weeks, in addition to a low-intensity psychosocial intervention program, with 26-week and 52-week follow-up observations.
  Baclofen: Baclofen 50mg per day for 12 weeks
- Placebo: Placebo, identical to baclofen was administered to the placebo group for 12 weeks
Period: Overall Study
Arm/Group | Baclofen | Placebo
Started | 32 | 32
Completed | 13 | 11
Not Completed | 19 | 21
Not completed — Lost to Follow-up | 10 | 16
Not completed — non compliance | 5 | 3
Not completed — condition worsened | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Patients were randomly assigned either to baclofen (N=32) or placebo (N=32) in a double-blind study design
- Total: Total of all reporting groups
Arm/Group | Baclofen | Placebo | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 24 | 24 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 32 | 32 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 32 | 32 | 64
Alcohol intake in last six months [Mean (Standard Deviation); unit: grams 40% alcohol/drinking day] | 763.6 (149.5) | 831 (151.0) | 797.3 (150.25)

OUTCOME MEASURES:

1. Primary Outcome: Percent Abstinent Days
Description: Percent abstinent days at 52 weeks. % of abstinent days were assessed by (1) patient's self-evaluation; (2) family member interview; (3) calculation of cumulative abstinence duration (CAD), defined as the total number of days of abstinence, Abstinent days was calculated for each Arm as a whole.
Time Frame: one year
Measure: Number; unit: percentage of abstinent days
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 13 | 11
percentage of abstinent days | 40 | 36

2. Secondary Outcome: Obsessive-Compulsive Drinking Scale Scores
Description: Used to evaluate self-reported alcohol craving. 14 items that provided a total (OCDS) as well as two subscale scores - obsessive drinking (OD) and compulsive drinking (CD). Each of the 14 items are scored from 0 to 4 with the inclusion of 4 split items with only the higher of the two scored items to be used in the total or subscale scores. The OCDS total score ranges from 0-40; the subscales both range from 0 to 20. On all scales, higher scores represent a worse outcome. Data for CD at 6 weeks not available to report
Time Frame: baseline, 6 weeks, 12 weeks, 26 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale
  OCDS at Baseline | 28.7 (9.8) | 28.6 (12.3)
  OD at Baseline | 11.4 (4.8) | 11.1 (5.1)
  CD at Baseline | 17.3 (6.8) | 17.6 (7.7)
  OCDS at 6 weeks (n=21,26) | 17.4 (9.2) | 15.1 (9.4)
  OD at 6 weeks (n=21,26) | 6.9 (4.3) | 6.1 (3.8)
  OCDS at 12 weeks (n=17,23) | 11.5 (9.3) | 12.8 (11.2)
  OD at 12 weeks (n=17,23) | 4.5 (3.9) | 4.6 (4.3)
  CD at 12 weeks (n=17,23) | 7.1 (5.9) | 8.3 (7.2)
  OCDS at 26 weeks (n=16,17) | 11.1 (10.1) | 7.9 (8.6)
  OD at 26 weeks (n=16,17) | 4.6 (4.3) | 3.4 (3.3)
  CD at 26 weeks (n=16,17) | 6.5 (6.6) | 4.3 (5.5)
  OCDS at 52 weeks (n=13,12) | 10.5 (10.1) | 7.8 (8.7)
  OD at 52 weeks (n=13,12) | 4.3 (4.1) | 3.4 (3.4)
  CD at 52 weeks (n=13,12) | 6.2 (6.9) | 3.6 (5.4)

3. Secondary Outcome: General Health Questionnaire
Description: The General Health Questionnaire measures whether the respondent has recently experienced a particular symptom or behavior and ranges from 0-much less than usual to 3-much more than usual. Total scores range from 0 to 36 and vary by study population: total scores of about 11-12 are typical, and a score higher than 20 suggests severe problems and psychological distress.
Time Frame: baseline, 6 weeks, 12 weeks, 26 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale
  Baseline | 17.7 (5.7) | 18.0 (6.2)
  Week 6 (n=21,26) | 15.1 (5.1) | 14.3 (5.9)
  Week 12 (n=17,23) | 13.2 (5.2) | 15.8 (7.1)
  Week 26 (n=16,17) | 9.9 (7.1) | 9.8 (12.5)
  Week 52 (n=13,12) | 10.1 (9.2) | 7.2 (7.9)

4. Secondary Outcome: General Self-Efficacy Scale
Description: The GSES measures one's belief in his/her ability to cope with stressful situations. The scale consists of 10 items (e.g. "Usually I am able to control a situation" or "In unexpected situations, I always know how I must behave myself"). Responses are rated on a 4- point Likert-scale ranging from "absolutely not true" (weighted as 1) to "absolutely true" (weighted as 4), where the higher GSES total scores indicate stronger self-efficacy beliefs.All responses are added to a sum score. The range is from 10 to 40 points with a higher score indicating more self-efficiency.
Time Frame: baseline, 6 weeks, 12 weeks, 26 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale
  Baseline | 25.4 (6.9) | 23.6 (8.3)
  Week 6 (n=21,26) | 24.1 (5.8) | 23.6 (6.6)
  Week 12 (n=17,23) | 27.8 (6.9) | 25.6 (6.0)
  Week 26 (n=16,17) | 27.1 (7.2) | 27.4 (6.9)
  Week 52 (n=13,12) | 25.8 (5.3) | 26.5 (6.0)

5. Secondary Outcome: Multidimensional Scale of Perceived Social Support
Description: The MSPSS is a self-report instrument for assessment of emotional help and the level of satisfaction with the social support obtained from three sources - family, friends and significant others. The scale includes 12 items, each of which refer to the people to whom the respondent would turn if he/she had problems of a personal, health or family nature, as well as financial and employment problems. Responses are scored on a 7-point scale from 1 ('completely disagree') to 7 ('completely agree'). The MSPSS index and three subscales - family, friends and significant others - are computed. MSPSS total score ranged from 12 to 84, with a higher score indicating greater satisfaction with total support. Subscores ranged from 4 to 28, with higher score indicating greater satisfaction.
Time Frame: Baseline, 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale
  Total at Baseline | 55.1 (18.3) | 55.2 (14.8)
  Family at Baseline | 19.4 (5.9) | 18.2 (6.7)
  Friends at Baseline | 15.6 (8.3) | 16.8 (6.6)
  Others at Baseline | 20.1 (7.0) | 20.3 (5.7)
  Total at 52 weeks (n=13,12) | 60.9 (18.7) | 55.9 (18.1)
  Family at 52 weeks (n=13,12) | 20.6 (6.3) | 18.3 (6.8)
  Friends at 52 weeks (n=13,12) | 18.3 (7.6) | 18.2 (5.5)
  Others at 52 weeks (n=13,12) | 20.8 (6.3) | 19.2 (7.0)

6. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q)
Description: Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) is a self-report form composed of 16 items, each rated on a 5-point scale that indicates the degree of enjoyment or satisfaction with: physical health; social relations; ability to function in daily life; ability to get around physically; mood; family relations; sexual drive and interest; ability to work on hobbies, work, leisure time activities; economic status; household activities; and living/housing situation. A total score of 1 to 15 items was computed while item 16 assessing "overall life satisfaction" was not included to avoid exaggerated scores. The total score was averaged from items 1 to 15 and ranged from 1 to 5, with higher scores indicating higher satisfaction.
Time Frame: baseline, 6 weeks, 12 weeks, 26 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: IThe placebo group received a placebo, identical to the baclofen medication for 12 weeks, in addition to a low-intensity psychosocial intervention program, with 26-week and 52-week follow-up observations
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale
  Baseline | 2.8 (0.8) | 2.8 (1.0)
  Week 6 (n=21,26) | 3.1 (0.8) | 3.2 (0.9)
  Week 12 (n=17,23) | 3.4 (0.7) | 3.4 (0.8)
  Week 26 (n=16,17) | 3.4 (0.6) | 3.6 (0.9)
  Week 52 (n=13,12) | 3.4 (0.8) | 3.6 (0.7)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Placebo: The placebo group received a placebo, identical to the baclofen medication for 12 weeks, in addition to a low-intensity psychosocial intervention program, with 26-week and 52-week follow-up observations.
Arm/Group | Baclofen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No